CLINICAL TRIAL: NCT00000551
Title: Activity Counseling Trial (ACT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 95
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

INTERVENTIONS:
Behavioral: health education

SUMMARY:
To develop and evaluate the effectiveness of various intervention approaches, delivered in primary health-care settings, in increasing and maintaining habitual physical activity and cardiorespiratory fitness among sedentary men and women patients.

DETAILED DESCRIPTION:
BACKGROUND:

A conference on physical activity sponsored by the National Heart, Lung, and Blood Institute (NHLBI) in August 1991 recommended that one priority area for research should be the development and evaluation of interventions for adoption and maintenance of physical activity including interventions that can be incorporated into primary care practice. The 1992 NHLBI Working Group Report on Primary Prevention of Hypertension identified physical inactivity as a risk factor for hypertension. Intervention research applicable to health-care settings is particularly important in light of national recommendations advising health-care professionals to intervene, including Healthy People 2000, the U.S. Preventive Services Task Force reports, and the American Heart Association.

DESIGN NARRATIVE:

Randomized, multicenter, demonstration and education study. Men and women primary care patients at three sites in Dallas, Palo Alto, and Memphis were randomized to two patient education intervention groups or to a standard care control group of physician advice. Intervention continued for two years for all participants. The primary outcomes were cardiorespiratory fitness and physical activity. Other outcomes were effects on blood pressure, lipoproteins, and weight; the long-term maintenance of these effects; and the cost-effectiveness of various intervention approaches. Recruitment took 15 months and has been completed with the accrual of 874 subjects.

The National Institute on Aging participated in the ACT through the addition of a measurement of arterial stiffness involving approximately 700 patients. The NIA tested the hypothesis that increases in physical activity resulting from educational interventions could reduce arterial stiffness.

ELIGIBILITY:
Sedentary men and women, free of coronary heart disease, who were patients in primary care settings.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-09; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgan — Bowman Gray School of Medicine

REFERENCES:
- [Background] King AC, Sallis JF, Dunn AL, Simons-Morton DG, Albright CA, Cohen S, Rejeski WJ, Marcus BH, Coday MC. Overview of the Activity Counseling Trial (ACT) intervention for promoting physical activity in primary health care settings. Activity Counseling Trial Research Group. Med Sci Sports Exerc. 1998 Jul;30(7):1086-96. doi: 10.1097/00005768-199807000-00011. PMID 9662678
- [Background] Simons-Morton DG. The context of the Activity Counseling Trial. Med Sci Sports Exerc. 1998 Jul;30(7):1084-5. doi: 10.1097/00005768-199807000-00010. No abstract available. PMID 9662677
- [Background] Blair SN, Applegate WB, Dunn AL, Ettinger WH, Haskell WL, King AC, Morgan TM, Shih JA, Simons-Morton DG. Activity Counseling Trial (ACT): rationale, design, and methods. Activity Counseling Trial Research Group. Med Sci Sports Exerc. 1998 Jul;30(7):1097-106. doi: 10.1097/00005768-199807000-00012. PMID 9662679
- [Background] Margitic S, Sevick MA, Miller M, Albright C, Banton J, Callahan K, Garcia M, Gibbons L, Levine BJ, Anderson R, Ettinger W. Challenges faced in recruiting patients from primary care practices into a physical activity intervention trial. Activity Counseling Trial Research Group. Prev Med. 1999 Oct;29(4):277-86. doi: 10.1006/pmed.1999.0543. PMID 10547053
- [Background] Havlik RJ, Brock D, Lohman K, Haskell W, Snell P, O'Toole M, Ribisl P, Vaitkevicius P, Spurgeon HA, Lakatta EG, Pullen P. High-density lipoprotein cholesterol and vascular stiffness at baseline in the activity counseling trial. Am J Cardiol. 2001 Jan 1;87(1):104-7, A9. doi: 10.1016/s0002-9149(00)01282-0. PMID 11137844
- [Background] Albright CL, Cohen S, Gibbons L, Miller S, Marcus B, Sallis J, Imai K, Jernick J, Simons-Morton DG. Incorporating physical activity advice into primary care: physician-delivered advice within the activity counseling trial. Am J Prev Med. 2000 Apr;18(3):225-34. doi: 10.1016/s0749-3797(99)00155-5. PMID 10722989
- [Background] Simons-Morton DG, Hogan P, Dunn AL, Pruitt L, King AC, Levine BD, Miller ST. Characteristics of inactive primary care patients: baseline data from the activity counseling trial. For the Activity Counseling Trial Research Group. Prev Med. 2000 Nov;31(5):513-21. doi: 10.1006/pmed.2000.0733. PMID 11071831
- [Background] Wee CC. Physical activity counseling in primary care: the challenge of effecting behavioral change. JAMA. 2001 Aug 8;286(6):717-9. doi: 10.1001/jama.286.6.717. No abstract available. PMID 11495623
- [Background] Havlik RJ, Phillips CL, Brock DB, Lohman K, Haskell W, Snell P, O'Toole M, Ribisl P, Vaitkevicius P, Spurgeon HA, Lakatta EG, Pullen P. Walking may be related to less vascular stiffness in the Activity Counseling Trial (ACT). Am Heart J. 2005 Aug;150(2):270-5. doi: 10.1016/j.ahj.2004.09.006. PMID 16086929
- [Background] Writing Group for the Activity Counseling Trial Research Group. Effects of physical activity counseling in primary care: the Activity Counseling Trial: a randomized controlled trial. JAMA. 2001 Aug 8;286(6):677-87. doi: 10.1001/jama.286.6.677. PMID 11495617
- Available data/document: Individual Participant Data Set: ACT — http://biolincc.nhlbi.nih.gov/studies/act/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/act/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/act/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/act/